CLINICAL TRIAL: NCT02198729
Title: Endoscopic Submucosal Dissection Versus Endoscopic Mucosal Resection for Sessile Polyps and Laterally Spreading Lesions of the Rectum - a Prospective Randomised Trial
Brief Title: Comparison Rectal Endoscopic Submucosal Dissection to Endoscopic Mucosal Resection
Acronym: RESDEMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC2013/10/4.2(3830)
Record Dates: First submitted 2014-07-17; First posted 2014-07-24 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endoscopic Mucosal Resection (Active Comparator): Participants randomised to this arm will receive standard of care Endoscopic Mucosal Resection for removal of their lesions.
  Interventions: Procedure: Endoscopic Mucosal Resection
- Endoscopic Submucosal Dissection (Experimental): Participants randomised to this arm will receive Endoscopic Mucosal Dissection to remove their lesion.
  Interventions: Procedure: Endoscopic Submucosal Dissection

INTERVENTIONS:
Procedure: Endoscopic Submucosal Dissection
  Arms: Endoscopic Submucosal Dissection
Procedure: Endoscopic Mucosal Resection
  Arms: Endoscopic Mucosal Resection

SUMMARY:
The investigators have recently become proficient in a new, and we believe more effective technique for polyp removal. Known as Endoscopic Submucosal Dissection (ESD). ESD involves removing the polyp in one piece. It is preferable to remove the polyp in one piece as it minimises the chance of leaving residual polyp tissue behind. There have also been recent studies overseas that have shown this new technique to be quite effective. In this study, half of the patients will receive the newly developed technique of polyp removal (ESD), while the other half will receive conventional Endoscopic Mucosal Resection (EMR) treatment. This study will allow us to show which technique results in lower recurrence rates and is more effective.

DETAILED DESCRIPTION:
EMR is a very effective procedure for lesions smaller than 20 mm. With this size the polyp can be removed en bloc. En bloc resection is preferred as it minimises the likelihood of residual adenoma and enhances histological assessment. It is also curative in superficially invasive submucosal disease. It eliminates the need for surgery in these patients. With lesions larger than 20 mm, the lesion is removed piece meal, often in more than 5 pieces. Care is taken to ensure that no adenoma is left behind at the point of overlap between snare resections. However, for every additional snare resection, there is the possibility that a small amount of adenoma will be left behind at this overlap point. Overall, the literature suggests that there is approximately a 15% residual adenoma rate at repeat colonoscopy in 3 months, which requires further treatment. With en bloc resection residual adenoma rate at repeat colonoscopy in is close to 0%. This has to be balanced against the relative inexperience with performing ESD, longer procedure time and higher complication rates. A randomized trial near completion is comparing endoscopic snare resection with transanal surgical resection for rectal polyps (24). Should this trial show that en bloc resection is superior in achieving complete resection without recurrence at similar complication rates, the endoscopic treatment strategy of large colorectal adenomas should be reconsidered. Since en bloc resection is technically more challenging, this should have consequences for credentialing, referral patterns and performance of removal of large colorectal polyps in reference centers only. Thus, before en bloc resection is promoted as superior, and training has to be intensified to comply with standards of safe oncologic resection of these lesions, the efficacy and safety have to be proven in a comparative randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Can give informed consent to trial participation
* Lesion size 20 mm to 50 mm
* Laterally spreading or sessile polyp morphology

Exclusion Criteria:

* Previous resection or attempted resection of target adenoma lesion
* Endoscopic appearance of invasive malignancy
* Age less than 18 years
* Pregnancy
* Active Inflammatory colonic conditions (e.g. inflammatory bowel disease)
* Use of anticoagulant or antiplatelet agents other than aspirin less than 5 days prior to procedure
* American Society of Anesthesiology (ASA) Grade IV-V

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2014-07; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Recurrence | 18 months
  Recurrence rate - free of adenoma endoscopically and histologically on 2 subsequent examinations

SECONDARY OUTCOMES:
One piece resection rate | 14 days
  Rate of en bloc resection
Technical success of EMR | 14 days
  Rate of initial technical success
Recurrence | up to 3 years
  Recurrence tissue observed at follow up colonoscopies over a 3 year period
complication rates | 14 days
  Safety outcomes measured in the form of follow up phone calls.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, MBBS, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Endoscopy Unit, Westmead, New South Wales, Australia

REFERENCES:
- [Derived] O'Sullivan T, Tate D, Sidhu M, Gupta S, Elhindi J, Byth K, Cronin O, Whitfield A, Craciun A, Singh R, Brown G, Raftopoulos S, Hourigan L, Moss A, Klein A, Heitman S, Williams S, Lee E, Burgess NG, Bourke MJ. The Surface Morphology of Large Nonpedunculated Colonic Polyps Predicts Synchronous Large Lesions. Clin Gastroenterol Hepatol. 2023 Aug;21(9):2270-2277.e1. doi: 10.1016/j.cgh.2023.01.034. Epub 2023 Feb 12. PMID 36787836